CLINICAL TRIAL: NCT06099327
Title: Image-based Remote Monitoring in Cardiac Surgery Patients: FORSEE 3 Trial
Brief Title: Image-based Remote Monitoring in Cardiac Surgery Patients
Acronym: FORSEE-3
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, Lukas Dekker, Prof. dr., Catharina Ziekenhuis Eindhoven
Other Study IDs: CZE-2023.28
Record Dates: First submitted 2023-09-12; First posted 2023-10-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Vital Signs; Clinical Deterioration
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Postoperative after cardiac surgery: Patients after cardiac surgery will participate in the trial during their postoperative stay on the cardiothoracic ward.
  Interventions: Device: Image-based vital sign monitoring

INTERVENTIONS:
Device: Image-based vital sign monitoring — Unobtrusive, vital signs measurements with remote photoplethysmography

SUMMARY:
In this observational study, 100 patients admitted to the Cardiothoracic ward will be additionally monitored with video-cameras. The video-cameras will measure heart- and respiration rate continuously. Other features, such a cardiac arrhythmias and context analysis may be added as well. Data will be analysed retrospectively and will be compared with vital parameters measured with healthdot- and spot check measurements.

DETAILED DESCRIPTION:
Rationale: In hospitals forty percent of unanticipated deaths occur in low-acuity departments. This alarming figure reflects the limited degree to which the cardiorespiratory status of patients is monitored in these departments, due to the obtrusiveness and expense of existing monitoring technologies, as well as the unpractically high clinical workload and costs that deployment of such technologies would entail. We have previously shown that an image-based monitoring technology reliably estimates heart rhythm and breathing rate under controlled conditions.

Objective: This project explores image-based monitoring of the cardiorespiratory status of patients as an innovative unobtrusive method that could eventually aid to reduce workload for the staff and better predict (acute) deterioration or adverse events. The purpose of this study is to evaluate the feasibility, in terms of system fidelity and acceptance, of long-term image-based monitoring in a cardiothoracic ward setting. Secondary objectives are to evaluate the validity of image-based vital signs and circadian rhythms in comparison with reference devices, the discriminative ability of image-based monitoring in the prediction of clinical deterioration and effect of clinical deterioration detected with remote monitoring during hospital admission on long-term patient outcomes.

Study design: Observational study Study population: 100 cardiac surgery patients

Main study parameters/endpoints: Primary endpoints are (1) insight in signal loss due to artifacts and time 'out of scope' of patients, (2) storage and processing solutions to enable conversion of large amounts of image-based data into vital signs and (3) level of acceptance by healthcare staff and patients. Secondary endpoints are performance of image-based vital signs and circadian rhythms in comparison with reference devices and sensitivity and specificity for the prediction of deterioration based on the image-based data. Moreover, potential time gain and predictive value of each image-based parameter will be assessed. Another secondary endpoint is insight in the relation of occurrence of clinical deterioration detected with the image-based monitoring technology during admission and long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing and able to sign informed consent form
* Patients admitted to the cardio-thoracic ward postoperative after cardiac surgery
* Planned stay on the cardio-thoracic ward at least 48 hours

Exclusion Criteria:

* Pregnant patients
* Inability to provide written informed consent
* Mental disability
* Language barrier
* Inability to wear Healthdot: known severe allergy for the tissue adhesive used in the Healthdot, any skin condition or use of topicals at the area of application of the Healthdot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population within this study will be cardiac surgery patients, admitted to the cardio-thoracic ward in the Catharina hospital, because they are at risk to develop postoperative complications. The research team will approach eligible patients who are scheduled to undergo cardiac surgery in collaboration with the cardio-thoracic surgeons. On average, 20 cardiac surgeries take place each week.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Percentage of signal coverage of remote, image-based monitoring in cardiac surgery patients on a general ward | 5-7 days
  Percentage of signal loss can be due to artifacts as a result movement, lighting conditions, clinical interventions and time 'out of scope' of patients

SECONDARY OUTCOMES:
The validity of remote, image-based heart- and respiration rate in comparison with heart- and respiration rate measured with the Healthdot (smart patch) | 5-7 days
  Agreement of image-based heart- and respiration rate with healthdot data
The validity of remote, image-based monitoring of circadian rhythms in comparison with the Healthdot (smart patch) | 5-7 days
  Agreement of image-based carcadian rhythms with healthdot data
Discriminative ability of remote, image-based monitoring in the detection of clinical deterioration | 1 year5-7 days
  Sensitivity/specificity of image-based data to predict clinical deterioration
Time to detection of clinical deterioration with the image-based monitoring technology vs conventional early warning score (measured via the spot check approach) | 5-7 days
  Potential time gain as a result of image-based monitoring in detection of clinical deterioration
Predictive value of each image-based parameter in the detection of postoperative complications | 5-7 days
  Added value of each image-based parameters in the detection of clinical deterioration
Effect of clinical deterioration detected with image-based, remote monitoring during hospital admission on long term patient outcomes (mortality, complications) | 2 years
  Association of occurence of postoperative complications with long term outcomes
Invasion of privacy of image-based remote monitoring, experienced by patients and healthcare staff, presented on a likert scale (1 means no invasion of privacy at all and 5 serious invasion of privacy) | 5-7 days
  Invasion of privacy will be assessed with a questionnaire with a likert scale (1-5), 1 means no invasion of privacy at all and 5 serious invasion of privacy.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Dekker, Prof. dr., Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided